CLINICAL TRIAL: NCT01670370
Title: A Prospective, Single-arm, Open-label, Phase 2 Study to Evaluate Efficacy and Safety of R-GemOx Regimen as First-line Treatment in Elderly Patients With Diffuse Large B-cell Lymphoma (DLBCL).
Brief Title: Trial of R-GemOx Regimen in Previously Untreated Elderly Patients With DLBCL.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-001
Record Dates: First submitted 2012-08-07; First posted 2012-08-22 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Rituximab; Gemcitabine; Oxaliplatin; Diffuse large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab+Gemcitabine+oxaliplatin (R-GemOx) (Experimental): Rituximab: 375 mg/m2 IV day1, Gemcitabine 1g/m2 IV day 2, oxaliplatin 100mg/m2 IV day2(every 14 days)
  Interventions: Drug: R-GemOx

INTERVENTIONS:
Drug: R-GemOx — Rituximab Gemcitabine Oxaliplatin
  Other Names: Rituximab; Gemcitabine; Oxaliplatin

SUMMARY:
The purpose of this study is to investigate efficacy and safety of GemOx(Gemcitabine and Oxaliplatin) combination with rituximab(R) as first-line treatment of elderly patients with DLBCL

DETAILED DESCRIPTION:
Previous studies showed that the combination of rituximab, gemcitabine and oxaliplatin (R-GemOx) achieved high efficacy with a low toxicity profile in relapsed and refractory DLBCL. This regimen might be considered a putative treatment option for elderly patients. To our knowledge, the efficacy and safety of R-GemOx when given as first-line therapy in elderly patients with DLBCL remains unknown. The investigators therefore developed a two-weekly regimen of rituximab combined with GemOx regimen as first line treatment in elderly DLBCL and investigate its efficacy and safety.

Primary Outcome Measures:

* overall response rate

Secondary Outcome Measures:

* progression free survival
* overall survival
* safety and toxicity

Enrollment: 60 Study Start Date: August 2012 Primary Completion Date: Dec 2015

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed CD20-positive DLBCL (The germinal center B-cell like (GCB) / non-GCB subtype was determined by immunohistochemistry in paraffin-embedded tissue using CD10, BCL6 and MUM1 protein markers based on Hans's algorithm);
2. New-diagnosed and untreated;
3. Age older than 70 years or older than 60 years with ECOG PS ≥2;
4. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Poor hepatic or renal function, defined as total serum bilirubin, transaminases or creatinine over two times of the upper limit of normal concentration;
2. Poor cardiac function greater than Grade II according to New York Heart Association Functional Classification;
3. Presence of Grade III nervous toxicity over two weeks;
4. Hepatitis B virus (HBV) load (HBV DNA) more than 1×105 copies/ml;
5. Concomitant malignancy other than DLBCL requiring treatment;
6. Concomitant with other hematologic diseases (such as leukemia, hemophilia, primary myelofibrosis) which is unsuitable to be enrolled into this clinical trial;
7. Contraindication to any drug in this regimen;
8. Active and severe infectious diseases, such as severe pheumonia or septicaemia;
9. Major surgery within three weeks;
10. Any medical, psychological or social conditions which might interfere with the investigators' assessment
11. In any conditions which investigator considered ineligible for this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | at the end of 3 cycles and 6 cycles of R-GemOx regimen(each cycle is 14 days)
  overall response rate after 3 cycles and at the end of R-GemOx regimen.

SECONDARY OUTCOMES:
progression free survival | Two-year
  from date of inclusion to date of progression, relapse from response, or death from any cause or last follow-up.
overall survival | Two-year
  from the date of inclusion to date of death, irrespective of cause or last follow-up.
The incidence and severity of adverse events | Up to 30 days following the last dose of study drug
  All the treatment related adverse events was evaluated according to common terminology criteria adverse events(CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: WEI XU, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

REFERENCES:
- [Background] Lopez A, Gutierrez A, Palacios A, Blancas I, Navarrete M, Morey M, Perello A, Alarcon J, Martinez J, Rodriguez J. GEMOX-R regimen is a highly effective salvage regimen in patients with refractory/relapsing diffuse large-cell lymphoma: a phase II study. Eur J Haematol. 2008 Feb;80(2):127-32. doi: 10.1111/j.1600-0609.2007.00996.x. Epub 2007 Nov 20. PMID 18005385
- [Background] Meriggi F, Zaniboni A. Gemox: a widely useful therapy against solid tumors-review and personal experience. J Chemother. 2010 Oct;22(5):298-303. doi: 10.1179/joc.2010.22.5.298. PMID 21123151
- [Derived] Shen QD, Zhu HY, Wang L, Fan L, Liang JH, Cao L, Wu W, Xia Y, Li JY, Xu W. Gemcitabine-oxaliplatin plus rituximab (R-GemOx) as first-line treatment in elderly patients with diffuse large B-cell lymphoma: a single-arm, open-label, phase 2 trial. Lancet Haematol. 2018 Jun;5(6):e261-e269. doi: 10.1016/S2352-3026(18)30054-1. Epub 2018 May 8. PMID 29752199